CLINICAL TRIAL: NCT02352428
Title: Skin Cancer Screening Education Study
Acronym: SCSES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association of Dermatological Prevention, Germany (Other)
Collaborators: University of Calgary (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LEO-SCSES_1013
Record Dates: First submitted 2015-01-13; First posted 2015-02-02 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Skin Tumors; Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Skin Cancer; Secondary Prevention; Population Screening
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin Cancer Screening Training (Experimental): Recruited family physicians and dermatologists in Calgary, Canada, take part in a 5.5-hour face-to-face skin cancer screening training program. Screening for skin cancer will be conducted by trained physicians according to instructions they received in the training program.
  Interventions: Other: Skin Cancer Screening Training
- No Skin Cancer Screening Training (No Intervention): Recruited family physicians and dermatologists in Edmonton, Canada, WILL BE TRAINED AFTER THE SCREENING PHASE, i.e. during the screening phase non-trained physicians will carry out skin cancer screenings according to standard medical practice.

INTERVENTIONS:
Other: Skin Cancer Screening Training — Topics of the 5.5-hour in-class course include: the screening test, types of skin cancer (signs and symptoms), case history taking, epidemiology of skin cancer, etiology, risk factors and risk groups, communicative aspects of primary and secondary preventive measures, and benefits and harms of cancer screenings.
  Arms: Skin Cancer Screening Training

SUMMARY:
The overall aim of this population-based screening study is to assess whether the skin cancer screening training of family physicians and dermatologists leads to improved screening outcomes. The training course aims to increase the accuracy of detecting early stages of skin cancer. Screening outcomes of an intervention region (Calgary, Canada) in which physicians receive training will be compared with screening outcomes of a control region (Edmonton, Canada) where no physician training is administered.

The investigators will determine whether:

* clinical screening outcomes are more favorable in the group of trained physicians compared to non trained physicians
* there is an increase of knowledge about skin cancer screening among trained physicians, compared to non trained physicians
* skin cancer screenings are associated with psycho-social harms
* population-based screening has an effect on the overall incidence and stage-specific-incidence of skin cancer in Alberta

The investigators are aiming to recruit 100 physicians per region (total of 200 physicians) who will screen 40,000 to 80,000 individuals over a period of 20 months.

ELIGIBILITY:
Inclusion Criteria:

1. Screenees

   * Male and female residents of Alberta mainly living and receiving care in Edmonton or in Calgary
   * Age 20+
   * English-speaking
   * Individuals who consent to participate
2. Physicians

   * Registered dermatologists and family physicians administering care either in Edmonton or in Calgary
   * English-speaking
   * Physicians who consent to participate

Exclusion Criteria:

Physicians who have undergone special training in skin cancer screening within the last 2 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in the diagnostic accuracy including knowledge on skin cancer screening | month 1 pre-training (intervention and control region), month 1 post-training (intervention region only), and month 12 (both regions)
  Educational outcomes of physicians will be measured pre- and post-training using knowledge tests in the intervention and control region
Number needed to screen (NNS) to identify 1 skin tumor and number needed to excise (NNE) to identify 1 skin tumor | 20 months
  Case report forms will be analyzed to determine clinical screening outcomes such as the NNS, NNE and tumor thickness.
Patient-rated well-being | 20 months
  A patient questionnaire will be used to assess psycho-social harms of skin cancer screenings.
Trends of overall skin cancer incidence and stage-specific-incidence | Up to 6 years (2012-2018)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Robertson, MD, FRCPC, Principal Investigator — University of Calgary; Gordon E Searles, MD, FRCPC, Principal Investigator — University of Alberta; Eckhard W Breitbart, MD, PhD, Principal Investigator — Association of Dermatological Prevention, Germany
Locations (1):
- University of Calgary, University of Alberta, Calgary, Edmonton, Alberta, Canada

REFERENCES:
- See also: Study website — http://www.scses-alberta.org